CLINICAL TRIAL: NCT03193541
Title: A Novel Multiplex ELISA Assay for Evaluating Patients With Microscopic Hematuria for Bladder Cancer
Status: Recruiting | Type: Observational
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Nonagen Bioscience Corporation (Industry); Nara Medical University (Other); University of California, Los Angeles (Other); University of Rochester (Other); National Cancer Institute (NCI) (NIH); University of Texas, Southwestern Medical Center at Dallas (Other); VA Long Beach Healthcare System (U.S. Federal Agency); Nara Prefecture Seiwa Medical Center (Unknown); University of Hawaii Cancer Research Center (Other); Fred Hutchinson Cancer Center (Other); Hoag Memorial Hospital Presbyterian (Other)
Responsible Party: Principal Investigator, Charles Rosser, Professor, Cedars-Sinai Medical Center
Other Study IDs: Rosser-2015-8; R01CA198887 (NIH)
Record Dates: First submitted 2017-06-17; First posted 2017-06-20 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine collection (minimal 50 mL) and cystoscopy (+ biopsy w/in 4 weeks, if abnormal noted)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To improve upon the non-invasive detection of BCa by further validating a multiplex ELISA assay directed at a BCa-associated diagnostic signature in voided urine samples of patients with microscopic hematuria.

DETAILED DESCRIPTION:
Hematuria is the most common presentation of BCa with 8% of patients with microscopic hematuria harboring BCa. VUC is the most widely used urine-based assay for detecting BCa; however, it fails to detect approximately 50% of low-grade or early stage BCa when it is most curable. Because of this severe limitation, patients with hematuria will undergo an invasive examination of the urinary bladder, where a miniature camera is inserted into the bladder.

We propose to improve the non-invasive detection of BCa by further validating a multiplex ELISA assay directed at a BCa-associated diagnostic signature in voided urine samples of patients with microscopic hematuria.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Have documented or reported microscopic hematuria within 3 month of study enrollment
* Willing and able to give written informed consent

Exclusion Criteria (participants must not):

* Have history of BCa
* History of previous cancer (excluding basal and squamous cell skin cancer)
* Have a known active urinary tract infection or urinary retention
* Have active stone disease (renal or bladder) or renal insufficiency (creatinine >2.0 mg/dL)
* Have ureteral stents, nephrostomy tubes or bowel interposition
* Have recent genitourinary instrumentation (within 10 days prior to signing consent)
* Be unable or unwilling to complete the hematuria evaluation (i.e., cystoscopy and upper tract imaging)

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults, age 18 and older who have documented microscopic hematuria within the past 3 months who are referred for cystoscopy and are willing to participate
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2016-12-30 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of multiplex ELISA assay will be confirmed by cystoscopy. | 1 year

SECONDARY OUTCOMES:
Sensitivity and specificity of multiplex ELISA assay will be compared to VUC and NMP-22 BladderChek. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Charles Rosser, MD, Study Director — Nonagen Bioscience Corporation; Hideki Furuya, PhD, Principal Investigator — Cedars-Sinai Medical Center
Locations (8):
- United States (6):
  - VA Long Beach Healthcare System, Long Beach, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - University of Rochester Medical Center, Rochester, New York
  - UT Southwestern Medical Center at Dallas, Dallas, Texas
- Japan (2):
  - Nara Prefecture Seiwa Medical Center, Nara, Nara
  - Nara Medical University, Nara

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Furuya H, Sakatani T, Tanaka S, Murakami K, Waldron RT, Hogrefe W, Rosser CJ. Bladder cancer risk stratification with the Oncuria 10-plex bead-based urinalysis assay using three different Luminex xMAP instrumentation platforms. J Transl Med. 2024 Jan 2;22(1):8. doi: 10.1186/s12967-023-04811-2. PMID 38167321
- [Derived] Furuya H, Sakatani T, Tanaka S, Murakami K, Waldron RT, Hogrefe W, Rosser CJ. Bladder cancer risk stratification with the Oncuria 10-plex bead-based urinalysis assay using three different Luminex xMAP instrumentation platforms. Res Sq [Preprint]. 2023 Nov 25:rs.3.rs-3635581. doi: 10.21203/rs.3.rs-3635581/v1. PMID 38045238